CLINICAL TRIAL: NCT03029767
Title: Effect of Aerobic and Resistance Exercise on Selected Anthropometric Biochemical and Physiological Variables Among Hypertensive Patients in Hawassa University Referral Hospital, Southern Ethiopia: a Parallel Randomized Controlled Trial
Brief Title: Effect of Exercise on Selected Anthropometric,Biochemical and Physiological Variables Among Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mekelle University (Other)
Responsible Party: Principal Investigator, Mitiku Daimo, Mitiku Daimo PhD scholar, Mekelle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213.55.94.37
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Hypertension
Keywords: Hypertension; Anthropometry; Aerobic exercise; Resistance exercise
MeSH Terms: conditions — Hypertension | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aerobic exercise (Experimental): Aerobic exercise training will be carried out as an intervention activity
  Interventions: Other: Aerobic exercise .
- Resistance exercise (Experimental): Resistance exercise training will be conducted as an intervention activity
  Interventions: Other: Resistance exercise
- Aerobic and resistance exercise (Experimental): Aerobic and resistance training will be implemented
  Interventions: Other: Aerobic and resistance exercise
- Control group (No Intervention): standard or usual activity carried out.Additional intervention will not be given.

INTERVENTIONS:
Other: Aerobic exercise . — The aerobic exercise group will perform brisk walking. Intensity of the aerobic exercise program will be progressively increased throughout the 16-week program. Intensity of aerobic exercise will be 40-65% of maximum heart rate , which is low to moderate.Duration of each session will be 45 minutes. Aerobic exercise will be performed 3 days per week.
  Other Names: Non pharmacological
  Arms: Aerobic exercise
Other: Resistance exercise — The resistance exercise group will perform 8 different exercises. Frequency of exercises per week is 3 days and duration of each exercise session is 45minutes. Interval rest among different exercises is 1minute.The intensity and repetition of resistance exercises is progressive. Participants will be exercised at 30% intensity (low intensity) for upper body and 50% intensity (moderate intensity) repetition voluntary maximum for lower body.
  Progressive, dynamic and rhythmical, alternative to upper-body and lower-body works and circuit resistance training of low to moderate intensity exercises will be executed.
  Other Names: Non pharmacological
  Arms: Resistance exercise
Other: Aerobic and resistance exercise — The aerobic and resistance exercise group will perform 23 minutes aerobic exercises and 22 minutes resistance exercises. The exercises will be performed three days per week . Intensity of aerobic and resistance exercise group for aerobic and resistance exercises are similar with intensity of aerobic group and resistance group exercises respectively.
  Other Names: Non pharmacological
  Arms: Aerobic and resistance exercise

SUMMARY:
Hypertension is the most common risk factor for development of stroke, congestive heart failure chronic kidney disease, and coronary artery disease in Sub Saharan Africa. The prevalence of hypertension will increase by 2025 in most parts of the world including Ethiopia according to World Health Organization.

Physical inactivity has been identified as a stronger predictor of chronic diseases such as hypertension. Exercise as a lifestyle modification is beneficial to a wide variety of health conditions, specific to hypertension; the benefits of exercise have been promoted by a number of organizations and agencies including World Health Organization.

According to the knowledge of the investigator there are no research works in relation to aerobic and resistance exercise effects among hypertensive patients generally in Ethiopia, and particularly in the area selected for the present research. Therefore the aim of this study is to assess the effect of aerobic and resistance exercises on selected anthropometric, biochemical and physiological variables among hypertensive patients in Hawassa University Referral Hospital.

DETAILED DESCRIPTION:
For eligible participants the requirements of the study will be explained and agree voluntarily to undergo the training and testing program. During orientation for each participant the risks, purpose, procedures and confidentiality of the requirement of the experiment testing as well as training protocol will be explained thoroughly prior to their written informed consent in their local language, and they have a full right to refuse from participating in this research or they have also the full right to withdraw from this study at any time they wish.

After acquisition of informed consent and exclusion criteria eligible participants will be randomized to one of four groups. Sequence allocation will be done by an individual who do not know and have no contact with the study participants .

Statistical analyses will be done using Statistical Package for Social Science (SPSS Version 20). One-way analyses of variance (ANOVA) will be used to assess differences between initial values of the four groups on all the variables measured. In addition, the effect of the experimental treatments on the anthropometric, biochemical and physiological variables will be examined by using two-way analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients who will give a written consent to participate in the study
* Hypertensive patients who are going to stay in the area throughout the study period
* Hypertensive patients between the age range of 31 and 45 years old with essential mild hypertension (systolic blood pressure between 140-159 mmHg and diastolic blood pressure between 90 and 99 mm Hg)
* participants not participated in structured physical exercises for previous 3 months
* patients who are on single anti-hypertensive medication or unmedicated
* Body mass index(BMI) 18.5kg/m2-29.9kg/m2

Exclusion Criteria:

* participants who involved in any exercise program prior to study
* pregnant women
* women who are taking contraceptive drugs
* Participants who are taking lipid lowering drugs
* participants who are taking any medications except single anti-hypertensive medication
* participants with organ damage,
* secondary hypertension
* patients with known liver problem
* patients with renal disease ,heart disease, brain disease
* participants with age less than 31 and greater than 45 years
* diabetic patients

Ages: 31 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-06-17 (Actual)

PRIMARY OUTCOMES:
Effect of aerobic exercise training (as intervention measures) on resting systolic blood pressure will be assessed. | [ Time Frame: sixteen weeks ]
  Change rates of systolic blood pressure among intervention and control groups

SECONDARY OUTCOMES:
Effect of combined aerobic and resistance training on the reduction of body mass index among the hypertensive patients will be assessed | [ Time Frame: Sixteen weeks ]
  Body mass index reduction changes among intervention and control groups
Effect of combined aerobic and resistance training on the increasement of HDL-c level among the hypertensive patients will be assessed | [ Time Frame: Sixteen weeks ]
  HDL-C level changes among intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Mitiku D Abebe, MSc, Principal Investigator — College of Natural and Computational Sciences,Mekelle University Mekelle University; Soumatra K Mondal, PhD, Study Director — College of Natural and Computational Sciences, Mekelle University Mekelle University; Mahmud Ab Mahmud, PhD, Study Chair — College of Health Sciences, Mekelle University; Palani B Kumar, PhD, Study Chair — College of Natural and Computational Sciences, Mekelle University
Locations (1):
- Hawassa University Referral Hospital, Awasa, Southern Nations Nationality Peoples Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Abstract of the study and consent format

REFERENCES:
- [Result] 1. Addo J, Smeeth L, Leon DA. Hypertension in sub Saharan Africa: a systematic review. Hypertension. 50(6):1012-8,2007. [PubMed/17954720] 2. Bacon SL, Sherwood A, Hinderliter A, Blumenthal JA. Effects of exercise, diet and weight loss on high blood pressure. Sports Medicine 35 (5), 307-316,2004. [PubMed/15107009] 3. Banz W, Maher M, Thompson W. Effects of resistance versus aerobic training on coronary artery disease risk factors. Exp Biol Med. 228(4):434-40,2003. [PubMed/12671188] 4. Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL, Jone JR, Materson BJ, Oparil S, Wright JT, Roccella EJ. Seventh Report of the Joint National Committee on prevention, detection, evaluation, and treatment of high blood pressure: the JNC 7 report.JAMA 289 (19):2560-72, 2003. [PubMed/12748199] 5. Cornelissen V, Fagard R. Effect of resistance training on resting blood pressure: a meta- analysis of randomized controlled trials. J Hypertens 23(2):251-9, 2005. [PubMed/15662209] 6. Cornelissen V, Fagard R. Effects of endurance training on blood pressure, blood pressure-regulating mechanisms, and cardiovascular risk factors. Hypertension 46 (4):667-75, 2005[PubMed/16157788] 7. Fagard RH, Cornelissen VA. Effect of exercise on blood pressure control in Hypertensive patients. Eur J Cardiovasc Prev Rehabil. 14:12-7, 2007. [PubMed/17301622] 8. Fagard RH. Exercise characteristics and the blood pressure response to dynamic physical training. Med Sci Sports Exerc 33: S484-492,2001. [PubMed/11427774] 9. Guidry, M.A., Blanchard ,B.E., Thompson ,P.D., Maresh, C.M., Seip, R.L., &Taylor, A.L. (2006). The influence of short and long duration on the blood pressure response to an acute bout of dynamic exercise. Am Heart J 151:1322.e5-12. [PubMed/16781245] 10. World Health Organization . Obesity: Preventing and Managing the Global Epidemic. WHO Technical Report 2000( 894). Geneva. 11. World Health Organization (2002). The world health report 2002: reducing risks, promoting healthy life. WHO, Geneva. 12. World Health Organization . The world health report 2002: reducing risks, promoting healthy life. WHO, Geneva 2000. 13. World Health Organization (WHO). A global brief on hypertension world health day. Geneva 2013. 14. Ha CH, So WY. Effects of combined exercise training on body composition and metabolic syndrome factors. Iran J Public Health. 41 (8):20-6,2012.[ PMC3469031]